CLINICAL TRIAL: NCT00962208
Title: Orthokeratology for Myopic Control in Chinese Children - a Randomized Clinical Trial
Brief Title: Retardation of Myopia in Orthokeratology
Acronym: ROMIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Menicon Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-ZG13
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2013-09-20 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-07

CONDITIONS: Myopia
Keywords: children; corneal reshaping; myopia; myopia control; orthokeratology
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- orthokeratology lenses (Experimental): Children wearing orthokeratology at night for correcting of refractive error will be study group
  Interventions: Device: orthokeratology lenses
- single-vision spectacle lenses (Other): Children wearing single-vision spectacles in the daytime for correcting the refractive error will serve as control group
  Interventions: Device: single-vision spectacle lenses

INTERVENTIONS:
Device: orthokeratology lenses — Nightly use of orthokeratology to correct the refractive error for a period of two years
  Other Names: Corneal reshaping therapy; Menicon Z Night Lens
  Arms: orthokeratology lenses
Device: single-vision spectacle lenses — Daily use of spectacles to correct the refractive error for a period of two years
  Other Names: CR-39 lenses
  Arms: single-vision spectacle lenses

SUMMARY:
The primary aim of this study is to evaluate and compare the eyeball elongation in children wearing orthokeratology lenses and single-vision spectacles.

DETAILED DESCRIPTION:
Prevalence of myopia is high in Asian countries like Hong Kong. Orthokeratology has shown potential in slowing myopic progression but the efficacy is yet to be confirmed by a randomized clinical trial (RCT). The current RCT aims at studying the efficacy of orthokeratology in retardation of myopic progression by comparing the eye growth in terms of axial length elongation in children wearing orthokeratology lenses (study group) and those wearing single-vision spectacles (control group).

ELIGIBILITY:
Inclusion Criteria:

* Myopia (refractive sphere): > 0.50D and ≤ 4.00D
* Astigmatism: < ½ of myopia; with-the-rule astigmatism (axes 180 +/- 30) ≤1.25D; astigmatism of other axes ≤ 0.50D
* Spherical equivalent (SE): > 0.75D and ≤ 4.50D
* Anisometropia: ≤ 1.50D in both refractive sphere, refractive cylinder and SE
* Best corrected monocular visual acuity: equal to or better than 0.10 in logMAR scale in both eyes
* Willingness for randomization
* Willingness to wear contact lenses or spectacles on a daily basis
* Availability for follow-up for at least 2 years

Exclusion Criteria:

* Strabismus at distance or near
* Contraindication for contact lens wear and orthokeratology (e.g. limbus to limbus corneal cylinder and dislocated corneal apex
* Prior experience with the use of rigid lenses (including orthokeratology)
* Prior experience with myopia control treatment (e.g. refractive therapy or progressive add spectacles)
* Systemic or ocular conditions which may affect contact lens wear (e.g. allergy and medication)
* Systemic or ocular conditions which may affect refractive development (e.g. Down syndrome, ptosis)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2008-03; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Background] Walline JJ, Jones LA, Sinnott LT. Corneal reshaping and myopia progression. Br J Ophthalmol. 2009 Sep;93(9):1181-5. doi: 10.1136/bjo.2008.151365. Epub 2009 May 4. PMID 19416935
- [Result] Cho P, Cheung SW. Retardation of myopia in Orthokeratology (ROMIO) study: a 2-year randomized clinical trial. Invest Ophthalmol Vis Sci. 2012 Oct 11;53(11):7077-85. doi: 10.1167/iovs.12-10565. PMID 22969068
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- [Derived] Cheung SW, Cho P. Validity of axial length measurements for monitoring myopic progression in orthokeratology. Invest Ophthalmol Vis Sci. 2013 Mar 5;54(3):1613-5. doi: 10.1167/iovs.12-10434. PMID 23361504
- [Derived] Chan KY, Cheung SW, Cho P. Clinical performance of an orthokeratology lens fitted with the aid of a computer software in Chinese children. Cont Lens Anterior Eye. 2012 Aug;35(4):180-4. doi: 10.1016/j.clae.2012.01.004. Epub 2012 Mar 3. PMID 22390958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phone screening was conducted on all parents who responded to advertisements in local newspapers during March 2008 and June 2009. Those who passed the screening would be invited to attend the baseline visit at the Optometry Clinic of The Hong Kong Polytechnic University.
Pre-assignment Details: All subjects who passed the inclusion and exclusion criteria at the baseline visit would be assigend to the treatment according to the randomization log.
Groups:
- Orthokeratology Lenses: Study group: children were asked to wear orthokeratology lenses every night (Menicon Z Night Lens: Menicon Z material, DK 163 ISO; central lens thickness: 0.24 mm) to correct the refractive error during the study period.
- Single-vision Spectacle Lenses: Control group: children were asked to wear single-vision spectacles (CR-39 material with refractive index 1.56) in the daytime to correct the refractive error during the study period.
Period: Overall Study
Arm/Group | Orthokeratology Lenses | Single-vision Spectacle Lenses
Started | 51 | 51
Completed | 37 | 41
Not Completed | 14 | 10
Not completed — Could not achieve good vision | 9 | 0
Not completed — Contraindicated to continue study | 5 | 1
Not completed — Lost to Follow-up | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Orthokeratology Lenses | Single-vision Spectacle Lenses | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 51 | 51 | 102
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.28 (1.10) | 9.27 (1.09) | 9.28 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 26 | 26 | 52
Region of Enrollment [Number; unit: participants]
  China | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Axial Elongation in the Study and Control Subjects Who Completed the Two Years Study
Description: Axial elongation was determined by the change in axial length of the eyeball before and after treatment period. Axial length was measured by the IOLMaster (Zeiss Humphrey, Dublin, CA) 30 minutes after cycloplegia. The measurement of the axial length followed the procedures as recommended by the manufacturer.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Orthokeratology Lenses | Single-vision Spectacle Lenses
Number analyzed (Participants) | 37 | 41
mm | 0.36 (0.24) | 0.63 (0.26)

2. Secondary Outcome: Determine the Incidence of Adverse Effects in Cornea, the Palpebral, Bulbar and Tarsal Conjunctiva in the Study and the Control Groups
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Determine Changes in Other Ocular Parameters (e.g. Corneal Biomechanics and Aberration) Associated With Orthokeratology Lens Wear
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Orthokeratology Lenses | Single-vision Spectacle Lenses
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes